CLINICAL TRIAL: NCT04928820
Title: Head-to-Head Comparison of 68Ga-PSMA-11 PET/CT With 99mTc-MDP Bone Scan and CT for Detection of M1b Disease in Prostate Cancer Patients With Biochemical Progression During ADT
Brief Title: 68Ga-PSMA-11 PET/CT for the Diagnosis of Bone Metastases in Patients With Prostate Cancer and Biochemical Progression During Androgen Deprivation Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-000102; NCI-2021-03575 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-10; First posted 2021-06-16 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Carcinoma; Stage IV Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (68Ga-PSMA-11 PET/CT) (Experimental): Patients receive gallium Ga 68 gozetotide IV. After 50-100 minutes, patients undergo whole body PET/CT.
  Interventions: Procedure: Computed Tomography; Other: Gallium Ga 68 Gozetotide; Procedure: Positron Emission Tomography

INTERVENTIONS:
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well 68Ga-PSMA-11 positron emission tomography (PET)/computed tomography (CT) works in detecting the spread of cancer to the bones (bone metastasis) in patients with prostate cancer and increased PSA after treatment (biochemical recurrence) during androgen deprivation therapy. Diagnostic procedures, such as 68Ga-PSMA-11 PET/CT, may help find and diagnose prostate cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the per-patient detection rate of 68Ga-PSMA-11 PET/CT versus bone scan (BS)/CT for M1b in patients treated with androgen deprivation therapy (ADT) who are referred for the imaging evaluation of disease progression.

SECONDARY OBJECTIVES:

I. To compare the number of lesions rated as positive for bone metastases between the two imaging tests.

II. To compare the detection rate of 68Ga-PSMA PET/CT versus BS/CT for all M1 disease (M1a or M1b or M1c).

III. To compare the positive predictive value (PPV) per-patient in patients with lesion validation (follow-up imaging or biopsy).

OUTLINE:

Patients receive gallium Ga 68 gozetotide intravenously (IV). After 50-100 minutes, patients undergo whole body PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Patient with biochemical progression during ADT or combination therapies including ADT who are referred for imaging evaluation (prostate specific antigen [PSA] level >= 1 ng/ml that has increased on at least 2 successive occasions at least 1 weak apart)
* Patients with bone scan scheduled or performed

  * Within 30 days of the PSMA PET, without any new prostate cancer (PCa) therapy in between
  * Bone scans performed at University of California, Los Angeles (UCLA) and external institutions are eligible if Digital Imaging and Communications in Medicine (DICOM) images can be obtained, imported, and anonymized
* Patients enrolled in other clinical trials are eligible if they satisfy all other criteria of eligibility
* Patients or their legal representatives must have the ability to read, understand and provide written informed consent

Exclusion Criteria:

* Initiation of a new therapy between the PSMA PET/CT and the bone scans
* Inability to provide written informed consent
* Known inability to remain still and lie flat for duration of each imaging procedure (about 30 minutes)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility requires prostrate gland
Enrollment: 22 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

PRIMARY OUTCOMES:
Per-patient detection rate of gallium Ga 68 gozetotide (68Ga-PSMA-11) positron emission tomography (PET)/computed tomography (CT) | Up to 4 years
  68Ga-PSMA-11 PET will be compared to bone scan/CT for M1b disease in prostate cancer patients progressing during androgen deprivation therapy. Patients who have at least one positive bone lesion will be rated positive. Patients will be treated as binary categorization. The analysis of the primary objective will utilize the McNemar's test to compare the detection rate between the imaging techniques.

SECONDARY OUTCOMES:
Number of lesions found by PSMA PET and bone scan + CT | Up to 4 years
  Will be compared using a paired samples t-test.
Rate of M1 detection | Up to 4 years
  Will be compared between the two modalities, defined as the number of patients with positive finding(s) for M1 disease (M1a or M1b or M1c), will utilize the McNemar's test for paired proportions.
Per-patient positive predictive value (PPV) | Up to 4 years
  Per-patient PPV estimates (with 95% confidence interval), defined as the number true positive findings the total number of positive cases (TP + FP). The lesions will be considered true positive on the basis of biopsy information, follow-up imaging, or changes in prostate specific antigen (PSA) levels. This information will only be available in a small subset of patients.
PSA progression-free survival (PFS) | Up to 4 years
  Univariate Cox proportional hazards models for PFS will be constructed with models containing various patient characteristics as well as PSMA PET parameters and bone scan parameters. Hazard ratios with 95% confidence intervals as well as p-values will be tabulated. Next, will explore multivariate models (using LASSO variable selection) including terms for important baseline characteristics as well as PSMA parameters or bone scan parameters and will extract the survival concordance indices from each of these models and compare them.
Overall survival (OS) | Up to 4 years
  Univariate Cox proportional hazards models for OS will be constructed with models containing various patient characteristics as well as PSMA PET parameters and bone scan parameters. Hazard ratios with 95% confidence intervals as well as p-values will be tabulated. Next, will explore multivariate models (using LASSO variable selection) including terms for important baseline characteristics as well as PSMA parameters or bone scan parameters and will extract the survival concordance indices from each of these models and compare them.
Incidence of adverse events | Up to 4 years
  Assessed using Common Terminology Criteria for Adverse Events version 4.03.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremie Calais, MD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- University of California at Los Angeles / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Nikitas J, Gafita A, Benz MR, Djaileb L, Farolfi A, Hotta M, Sonni I, Alano R, Rettig M, Shen J, Armstrong W, Grogan T, Liu S, Czernin J, Calais J. Phase 2 trial of PSMA PET CT versus planar bone scan and CT in prostate cancer patients progressing while on androgen deprivation therapy. Sci Rep. 2024 Oct 18;14(1):24411. doi: 10.1038/s41598-024-75589-6. PMID 39420060